CLINICAL TRIAL: NCT02271074
Title: An Evaluation of Strategies to Accelerate Entry-into-care Following HIV Diagnosis Among Adults in Gauteng and Limpopo Provinces, South Africa
Brief Title: Thol'Impilo: Bringing People Into Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AUR5-9-119; AID-OAA-A-12-00028 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2014-10-14; First posted 2014-10-22 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-01

CONDITIONS: HIV
Keywords: HIV; Care; Treatment; Retention; Implementation Science

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard of Care (No Intervention): The role of this arm is to provide a baseline measure that can be used to assess the effectiveness of the combination interventions in improving the proportion of individuals entering care within 3 months. Participants in this arm only receive standard post-test counselling after they are issued with a positive HIV result. They are counselled on possible emotional resources, and given information on how to reduce risk of HIV transmission, ongoing positive living, nutrition and healthy lifestyles. These clients are given referral letters and referred to health facilities of their choice that offer HIV care/treatment. They are then followed up at the designated study time points to ascertain entry into care.
- Point of care CD4 testing (Experimental): Participants in this arm will receive point of care (POC) cluster differentiation 4 (CD4) testing using the PIMA™ CD4 test system.
  Interventions: Other: Point of care CD4 testing
- Care facilitation (Experimental): Participants receive a combination of POC CD4 testing and care facilitation.
  Interventions: Other: Point of care CD4 testing; Behavioral: Care Facilitation
- Transport support (Experimental): Participants receive a combination of POC CD4 testing and transport support.
  Interventions: Other: Point of care CD4 testing; Other: Transport support

INTERVENTIONS:
Other: Point of care CD4 testing — Participants in this arm will receive POC CD4 testing using the PIMA™ CD4 test system. Results will be made available to the participant within 20 to 25 minutes, before the participant leaves the HCT room. Participants will be given a copy of their results, which will be affixed to their referral letter, and they will be educated on the meaning of the CD4 results in relation to their health. This session will only be performed once at the time of issuing POC CD4 results.
  Arms: Care facilitation; Point of care CD4 testing; Transport support
Behavioral: Care Facilitation — The goal of this intervention is to provide on-going counselling using a combination of motivational and strengths-based counselling approaches.This is a time limited intervention with a maximum of 5 client sessions over a 90-day period. Participants will also be transitioned out of the intervention upon successful entry into HIV care. Sessions will be done using both face-to-face and telephonic approaches, although the former is more preferred.
  Arms: Care facilitation
Other: Transport support — The goal of this intervention is to address one of the most frequently noted structural barrier to entry-into-care in resource constrained settings: prohibitive distance or transport cost to reach a health facility.This is a time limited intervention with a maximum of 3 transport assists for healthcare visits over a 90-day period. Transport assistance is provided in the form of reimbursements to claims submitted by the participant after a self-reported HIV care clinic visits. Participants in this arm, receive their transport support through in-person collection or via cell phone transfer. Transport support amounts are standardised according to geographical area.
  Arms: Transport support

SUMMARY:
The main objective of this study is to compare the effectiveness of combinations of three patient-oriented strategies, compared to the standard of care, to increase the proportion of patients who enter-into-care for HIV within 90 days of testing HIV positive.

DETAILED DESCRIPTION:
Background:

Mortality remains high among individuals with HIV in South Africa largely due to low CD4 at initiation of combination antiretroviral therapy (cART) or failure to initiate cART altogether. The problem of advanced HIV at the time of entry-into-care persists despite increases in CD4 count initiation thresholds and higher CD4 counts among individuals testing HIV positive at HIV counselling and testing services (HCT). A reason for the discord between CD4 at HCT and CD4 at cART initiation is a failure to effectively link people who test positive into HIV care; less than half of individuals testing HIV positive enter HIV care within 3-6 month of HIV diagnosis. However, not only do these delays increase HIV associated mortality, delays from testing positive to entry-into-care for HIV also reduces the ability of test-and-treat strategies to reduce HIV transmission through HIV treatment.

Study Design:

Thol'impilo is an open (non-masked) individually-randomized implementation science evaluation of the effectiveness and cost-effectiveness of combinations of three strategies to increase timely entry-into-care for HIV compared to the standard of care. Participants are randomly assigned to one of four arms to increase timely entry into care: (1) standard of care, (2) point-of-care CD4 and transport assistance, (3) point-of-care CD4 and care facilitator and (4) point-of-care CD4 alone.

Sample size:

The study aims to enrol 2500 participants (i.e. 650 participants per arm).

Setting:

The study is built onto the current community-based HIV Counselling and Testing (HCT) services. The HCT units serve peri-urban townships and informal settlements, rural farm workers, and both urban and rural communities.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older, diagnosed HIV positive at enrolling mobile HCT units, no prior self-reported registration at a health care facility for HIV care, provide consent for participation

Exclusion Criteria:

* self-reported prior or current registration as an HIV patient at a healthcare facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2398 (Actual)
Dates: Start 2012-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Time to entry into HIV care | 90 days
  To compare the time to entering HIV care in each intervention arm against the standard of care arm over a 90 day period from study enrolment.

SECONDARY OUTCOMES:
Proportion entering care | 90 days
  To compare the proportion of participants in each arm entering care by 90 days from study enrolment
Time to entry into HIV care | 180 days
  To compare the time to entering HIV care in each intervention arm against the standard of care over a 180 day period from study enrolment.
Mortality | 6 and 12 months
  To compare time to mortality from enrolment by arm over a 12 month period
Cost per additional participant entering into care | Costs will be measured over a 12 month horizon and entry into care will be measured over a 90 day period
  To evaluate the incremental cost effectiveness (cost per additional participant entering into care by 90 days) for each intervention arm compared to the standard-of-care

OTHER OUTCOMES:
Time to ART initiation | 90 days
  To compare the proportion of cART-eligible patients who initiate cART within 90 days of study enrolment in each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Violet Chihota, PhD, Study Director — The Aurum Institute NPC
Locations (1):
- The Aurum Institute NPC, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through identified USAID -PEPFAR Platforms.

REFERENCES:
- [Derived] Hoffmann CJ, Mabuto T, Ginindza S, Fielding KL, Kubeka G, Dowdy DW, Churchyard GJ, Charalambous S. Strategies to Accelerate HIV Care and Antiretroviral Therapy Initiation After HIV Diagnosis: A Randomized Trial. J Acquir Immune Defic Syndr. 2017 Aug 15;75(5):540-547. doi: 10.1097/QAI.0000000000001428. PMID 28471840